CLINICAL TRIAL: NCT01466114
Title: A Double-Blind, Placebo Controlled Trial of Estriol Treatment in Women With Multiple Sclerosis: Effect on Cognition.
Brief Title: Estriol Treatment in Multiple Sclerosis (MS): Effect on Cognition
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Rhonda Voskuhl, Professor, Department of Neurology; Director Multiple Sclerosis Program, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-002055
Record Dates: First submitted 2011-10-31; First posted 2011-11-07 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Relapsing-remitting Multiple Sclerosis; Secondary-progressive Multiple Sclerosis; Primary-progressive Multiple Sclerosis
Keywords: multiple sclerosis; MS; relapsing remitting multiple sclerosis; RRMS; secondary progressive multiple sclerosis; SPMS; primary progressive multiple sclerosis; estrogen; estriol
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — Estriol; estriol succinate; Norethindrone; Progestins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Estriol (Experimental): Standard MS Treatment + Estriol
  Interventions: Drug: estriol; Drug: Norethindrone
- Group B: Placebo (Placebo Comparator): Standard MS Treatment + Placebo
  Interventions: Other: Placebo; Other: Progestin Placebo

INTERVENTIONS:
Drug: estriol — 4 capsules of 2 mg (total of 8 mg) PO QD
  Other Names: Synapause
  Arms: Group A: Estriol
Other: Placebo — 4 capsules PO QD
  Arms: Group B: Placebo
Drug: Norethindrone — Starting at month 6, and at Months 9 and 12: subjects who are on estriol (Group A) take 0.7 mg PO QD for 2 weeks.
  Other Names: Progestin
  Arms: Group A: Estriol
Other: Progestin Placebo — Starting at Month 6 and at Months 9 and 12: subjects who are on placebo (Group B) take a second progestin placebo pill PO QD for 2 weeks.
  Arms: Group B: Placebo

SUMMARY:
Approximately 50% of people diagnosed with Multiple Sclerosis (MS) will develop problems with cognition. Currently, there are no FDA-approved treatments targeting cognitive function in Multiple Sclerosis. This trial will ascertain whether treatment with an estrogen pill, used in combination with standard MS anti-inflammatory drugs, can improve cognitive testing as compared to treatment with a placebo pill in combination with standard anti-inflammatory drugs in women with MS.

DETAILED DESCRIPTION:
Approximately 50% of people diagnosed with Multiple Sclerosis (MS) will develop problems with cognition. Currently, there are no FDA-approved treatments for cognitive function in Multiple Sclerosis. Multiple sclerosis relapses are known to be significantly decreased by approximately 80% during late pregnancy. This disease improvement may be due to estriol, an estrogen unique to pregnancy. Estriol blood levels go from undetectable levels prior to pregnancy, increase during pregnancy and reach highest levels during late pregnancy. Further, estrogen treatment has been shown to have favorable effects on cognition in animal models of other neurological diseases. This proposal will establish whether oral treatment with estriol, induces an improvement in cognitive functioning in subjects with multiple sclerosis when used in combination with the major FDA-approved standard treatments for MS, (Betaseron® (or Extavia®), Rebif®, Avonex®, Copaxone®, Gilenya®, Aubagio®, Tecfidera®, or Ocrevus®).

The combination of standard MS treatment plus estriol pill (8 mg per day) will be compared to standard MS treatment plus placebo in a double-blinded fashion. The duration of treatment will be one year and the primary outcome measure will be cognitive testing processing speed ability.

Secondary outcomes will be improvement in other cognitive tests, brain MRIs, cognitive evoked potentials, as well as relapse rates and disability measures (EDSS, 25 foot walk, 9 hole peg test, low contrast visual acuity, MS Quality of Life, Modified Fatigue Impact Scale, Beck Depression Inventory, Level of Activity using accelerometry). Safety measures (blood tests and gynecologic evaluations) will also be followed. The overall goal of this study will be the development of an oral treatment, estriol, to improve cognitive function in MS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinically definite or MacDonald criteria relapsing-remitting multiple sclerosis, secondary-progressive multiple sclerosis or primary-progressive multiple sclerosis.
* No relapse within 30 days before day of trial enrollment (month 0 visit). If steroids given for relapse, then the month 0 visit must be 30 days after last steroid dose.
* Females age 18 to 55, inclusive.
* Expanded Disability Status Score (EDSS) = 0.0 to 6.0.
* Screening PASAT (3-second) score 25-50, inclusive.
* Must be mentally competent enough to comply with study guidelines and give informed consent.
* Must be willing and able to travel to the study center at frequencies in the protocol for a total period of 12 months.
* Patients must be on no treatment or be on a stable dose of one of the following agents for a minimum of 3 months duration prior to the month 0 visit: Copaxone®, Betaseron® (or Extavia®), Rebif®, Avonex®, PLEGRITY®, Ocrelizumab, Rituximab, Gilenya®, Aubagio®, or Tecfidera®. The time spent in the screening period may serve as part of this 3-month period.
* Patients who are currently being treated with ACTH, corticosteroids, intravenous immunoglobulins (IVIG), plasma exchange, Lipitor® or minocycline may be included.
* If patients plan to start treatment with Copaxone® or an interferon [Betaseron® (or Extavia®), Rebif®, Avonex®, PLEGRITY®], Ocrelizumab, Rituximabor an oral agent [Gilenya®, Aubagio® or Tecfidera®] and then they must be on for at least 3 months prior to month 0 (as above).

Exclusion Criteria:

* Males
* Subjects on oral contraceptives (OCP), hormone replacement therapy (HRT) other sex hormones during screening and during the 12-month study period (Mirena® IUD is permitted).
* Females who are pregnant or who plan to become pregnant during the 12 months of enrollment, who wish to become pregnant within 3 months following completion of the study, or who will be within 6 months post partum at the day of first enrollment visit (month 0).
* Females who plan to breastfeed after first enrollment visit (month 0).
* Fertile sexually active women who are unwilling to practice reliable barrier methods of contraception other than oral contraceptives (i.e. condom, diaphragm, IUDs Note: Hormonal IUD [Mirena®] is permitted).
* Patients with surgical ovariectomy with no hormone replacement for 1 year or more.
* Menopause with no hormone replacement for 3 years or more prior to the first enrollment visit.
* Patients who smoke at any time during screening or during the 12 month study period.
* Patients who have serious pulmonary, renal, gastrointestinal, hepatic, immunologic, infectious, neoplastic, major psychiatric disease (major depression, schizophrenia), endocrine disease (including major diabetes, thyroid disease), or gynecologic disease, including but not limited to those with: Thrombophlebitis or thromboembolic disorders, a past history of deep vein thrombophlebitis or thromboembolic disorders, cerebral vascular or coronary artery disease, migraine with focal aura, known or suspected carcinoma of the breast, carcinoma of the endometrium or other known or suspected estrogen-dependent neoplasia, undiagnosed abnormal genital bleeding, polycystic ovary disease, amenorrhea of unknown etiology, cholestatic jaundice of pregnancy or jaundice with prior birth control pill use, acute or chronic hepatocellular disease with abnormal liver function, hepatic adenomas or carcinomas, known or suspected pregnancy, known hypersensitivity to birth control pill Copaxone or Betaseron use.
* B12 level < 200.
* Drug abuse within the past five years.
* Conditions that would interfere with assessing neurologic functions such as deforming arthritis or a major amputation.
* Have at any time been treated with total lymphoid irradiation, monoclonal antibody, T cell vaccination, cladribine, bone marrow transplantation, azathioprine, cyclophosphamide, methotrexate, mitoxantrone, or cyclosporine.
* Have been treated with natalizumab (Tysabri®) in the 6 months prior to screening.
* Positive titers to HIV in the past.
* Previous serious adverse effects with estrogen treatment.
* Patients who participated in the previous multi-center estriol trial for RRMS ("A Combination Trial of Copaxone plus Estriol in RRMS").

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2011-10; Primary Completion 2021-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in cognitive function assessed by Paced Serial Addition Test (PASAT). | 1 year
  Processing speed will be assessed by PASAT. Numerical test scores (ranging from 0-60) will be acquired, then percent change for each subject at trial conclusion as compared to baseline will be determined. Whether greater improvement as expressed as percent change occurs in the estriol group as compared to the placebo group will be determined.

SECONDARY OUTCOMES:
Change from baseline in cognitive function as assessed by cognitive evoked potentials, measured in milliseconds. | 1 year
  Cognitive evoked potentials will be recorded in msecs for each subject at baseline and conclusion. The percent improvement as conclusion as compared to baseline for each subject will be determined. Group comparisons will reveal whether the percent improvement is greater in the estriol treated group as compared to the placebo treated group.
Change from baseline in standard MS outcome measures. | 1 year
  Determine whether the combination treatment has an effect on standard MS outcome measures (relapses, EDSS, 25 foot walk test, 9 hole peg test, low contrast visual acuity, MS Quality of Life, Modified Fatigue Impact Scare, Beck Depression Inventory.
Determine safety by assessing the number of subjects with adverse events with combination treatment as compared to placebo. | 1 year
  Determine whether the combination treatment is safe (based on neurologic exams, laboratory tests (Chemistries, CBC), and gynecologic exams (breast and gynecologic exams).
Change from baseline in cognitive function as assessed by a brief battery of cognitive tests. | 1 year
  A brief battery of cognitive tests will be administered including: Processing speed: SDMT-hand written; Visual memory: 7/24 Spatial Recall Test, Benton Forms F & G; Verbal memory: Buschke Selective Reminding Test, Verbal Paired Associates; Language: Word List Generation. Each subject will be tested at baseline, month 6 and conclusion. Percent change at conclusion as compared to baseline will be determined in each subject. Group comparisons will reveal which cognitive test within the battery had greater improvement in the estriol treated group as compared to the placebo treated group.

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Voskuhl, M.D., Principal Investigator — University of California, Los Angeles
Locations (4):
- United States (4):
  - University of California Los Angeles, Los Angeles, California
  - The University of Colorado Denver, Aurora, Colorado
  - The University of New Mexico, Albuquerque, New Mexico
  - The University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Ziehn MO, Avedisian AA, Dervin SM, O'Dell TJ, Voskuhl RR. Estriol preserves synaptic transmission in the hippocampus during autoimmune demyelinating disease. Lab Invest. 2012 Aug;92(8):1234-45. doi: 10.1038/labinvest.2012.76. Epub 2012 Apr 23. PMID 22525427
- [Background] Voskuhl RR, Wang H, Wu TC, Sicotte NL, Nakamura K, Kurth F, Itoh N, Bardens J, Bernard JT, Corboy JR, Cross AH, Dhib-Jalbut S, Ford CC, Frohman EM, Giesser B, Jacobs D, Kasper LH, Lynch S, Parry G, Racke MK, Reder AT, Rose J, Wingerchuk DM, MacKenzie-Graham AJ, Arnold DL, Tseng CH, Elashoff R. Estriol combined with glatiramer acetate for women with relapsing-remitting multiple sclerosis: a randomised, placebo-controlled, phase 2 trial. Lancet Neurol. 2016 Jan;15(1):35-46. doi: 10.1016/S1474-4422(15)00322-1. Epub 2015 Nov 29. PMID 26621682
- [Background] Voskuhl R, Wang H, Elashoff RM. Why use sex hormones in relapsing-remitting multiple sclerosis? - Authors' reply. Lancet Neurol. 2016 Jul;15(8):790-791. doi: 10.1016/S1474-4422(16)00129-0. No abstract available. PMID 27302354
- [Background] Voskuhl R, Patti F. Hormone replacement in menopausal women with multiple sclerosis: Looking back, thinking forward. Neurology. 2016 Oct 4;87(14):1430-1431. doi: 10.1212/WNL.0000000000003189. Epub 2016 Sep 7. No abstract available. PMID 27605172
- [Background] Voskuhl R. Rebound Relapses After Ceasing Another Disease-Modifying Treatment in Patients With Multiple Sclerosis: Are There Lessons to Be Learned? JAMA Neurol. 2016 Jul 1;73(7):775-6. doi: 10.1001/jamaneurol.2016.0934. No abstract available. PMID 27136400
- [Background] Itoh N, Kim R, Peng M, DiFilippo E, Johnsonbaugh H, MacKenzie-Graham A, Voskuhl RR. Bedside to bench to bedside research: Estrogen receptor beta ligand as a candidate neuroprotective treatment for multiple sclerosis. J Neuroimmunol. 2017 Mar 15;304:63-71. doi: 10.1016/j.jneuroim.2016.09.017. Epub 2016 Oct 3. PMID 27771018
- [Background] Kim RY, Mangu D, Hoffman AS, Kavosh R, Jung E, Itoh N, Voskuhl R. Oestrogen receptor &beta; ligand acts on CD11c&plus; cells to mediate protection in experimental autoimmune encephalomyelitis. Brain. 2018 Jan 1;141(1):132-147. doi: 10.1093/brain/awx315. PMID 29228214
- [Background] MacKenzie-Graham A, Brook J, Kurth F, Itoh Y, Meyer C, Montag MJ, Wang HJ, Elashoff R, Voskuhl RR. Estriol-mediated neuroprotection in multiple sclerosis localized by voxel-based morphometry. Brain Behav. 2018 Sep;8(9):e01086. doi: 10.1002/brb3.1086. Epub 2018 Aug 24. PMID 30144306
- [Background] Voskuhl RR, Itoh N, Tassoni A, Matsukawa MA, Ren E, Tse V, Jang E, Suen TT, Itoh Y. Gene expression in oligodendrocytes during remyelination reveals cholesterol homeostasis as a therapeutic target in multiple sclerosis. Proc Natl Acad Sci U S A. 2019 May 14;116(20):10130-10139. doi: 10.1073/pnas.1821306116. Epub 2019 Apr 30. PMID 31040210
- [Background] Voskuhl R. It is time to conduct phase 3 clinical trials of sex hormones in MS - Yes. Mult Scler. 2018 Oct;24(11):1413-1415. doi: 10.1177/1352458518768764. Epub 2018 Jul 30. No abstract available. PMID 30058469
- [Background] Voskuhl R, Momtazee C. Pregnancy: Effect on Multiple Sclerosis, Treatment Considerations, and Breastfeeding. Neurotherapeutics. 2017 Oct;14(4):974-984. doi: 10.1007/s13311-017-0562-7. PMID 28766273